CLINICAL TRIAL: NCT04157426
Title: Effectiveness of Ultrasound-guided Interventions of Percutaneous Electrolysis Versus Dry Needling in Levator Scapulae Active Myofascial Trigger Points
Brief Title: Percutaneous Electrolysis Versus Dry Needling in Levator Scapulae
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, César Calvo Lobo, Principal Investigator, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PE_vs_DN
Record Dates: First submitted 2019-11-06; First posted 2019-11-08 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Trigger Point Pain, Myofascial; Myofascial Pain
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-guided percutaneous electrolysis (Experimental)
  Interventions: Other: Percutaneous electrolysis
- ultrasound-guided dry needling (Active Comparator)
  Interventions: Other: Dry needling

INTERVENTIONS:
Other: Percutaneous electrolysis — Ultrasound-guided percutaneous electrolysis in the active myofascial trigger point of the levator scapulae muscle
  Arms: Ultrasound-guided percutaneous electrolysis
Other: Dry needling — Ultrasound-guided dry needling the active myofascial trigger point of the levator scapulae muscle
  Arms: ultrasound-guided dry needling

SUMMARY:
The objective will be to determine the effectiveness of ultrasound-guided percutaneous electrolysis versus ultrasound-guided dry needling in active myofascial trigger points of the levator scapulae muscle on pain intensity, disability and range of motion. A randomized clinical trial will be carried out. Fifty-four patients with at least one active myofascial trigger point in the levator scapulae muscle were recruited and divided into ultrasound-guided percutaneous electrolysis (n = 27) and ultrasound-guided dry needling (n=27). Pain intensity, disability and range of motion will measured before, immediately after and 1 week after intervention.

ELIGIBILITY:
Inclusion Criteria:

* Neck pain
* At least two active myofascial trigger point in the levator scapulae muscle

Exclusion Criteria:

* Systemic diseases
* Cognitive impairment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Change from baseline pain intensity immediately and at 1 week after intervention
  Neck pain intensity scores from 0 to 100 points measured by the visual analogue scale

SECONDARY OUTCOMES:
Disability | Change from baseline pain intensity at 1 week after intervention
  Neck disability scores measured from 0 to 50 points measured by the Neck Disability Index
Range of motion | Change from baseline pain intensity immediately and at 1 week after intervention
  Neck rotation range of motion measured with an universal goniometer

CONTACTS AND LOCATIONS:
Locations (1):
- Fisiofuenla SLP, Fuenlabrada, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Benito-de-Pedro AI, Becerro-de-Bengoa-Vallejo R, Losa-Iglesias ME, Rodriguez-Sanz D, Calvo-Lobo C, Benito-de-Pedro M. Efficacy of Deep Dry Needling versus Percutaneous Electrolysis in Ultrasound-Guided Treatment of Active Myofascial Trigger Points of the Levator Scapulae in Short-Term: A Randomized Controlled Trial. Life (Basel). 2023 Apr 3;13(4):939. doi: 10.3390/life13040939. PMID 37109468